CLINICAL TRIAL: NCT00498082
Title: Determinants of Efficacy of EsophyX Treatment in Gastro-Esophageal Reflux Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Other Study IDs: UCL-STLUC-GAS-01
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2007-09-06 (Estimated); Status verified 2007-09

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
EsophyX is a promising endoscopic treatment for gastro-esophageal reflux disease. It is not known whether there are some pre- or per-operative anatomic or pathophysiological findings which may influence outcome.

The aim of this trial is to study a series of parameters acquired during the pre-therapeutic work-up or during the procedure and their influence on the outcome of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients being considered for EsophyX treatment of GERD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-09; Study Completion 2008-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Piessevaux, MD, PhD, Principal Investigator — Cliniques universitaires St-Luc
Locations (1):
- Cliniques universitaires St-Luc, Brussels, Belgium

REFERENCES:
- See also: Cliniques universitaires St-Luc — http://www.saintluc.be